CLINICAL TRIAL: NCT06446895
Title: Biomarkers of Inflammation and Endothelial Dysfunction in Patients With Myocardial Infarction With Non-obstructive Coronary Arteries
Acronym: IMACORN-INFLI
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, maria jesus espinosa pascual, Cardiologist, Hospital Universitario Getafe
Other Study IDs: IMACORN-INFLI
Record Dates: First submitted 2024-05-27; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-05

CONDITIONS: Myocardial Infarction; MINOCA; Inflammation; Biomarkers; Endothelial Dysfunction
MeSH Terms: conditions — Myocardial Infarction; MINOCA; Inflammation | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, plasma, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MICAD: Patients with Myocardial Infarction and Obstructive Coronary Arteries
  Interventions: Diagnostic Test: Coronariography
- MINOCA: Patients with Myocardial Infarction and Non-obstructive Coronary Arteries
  Interventions: Diagnostic Test: Coronariography

INTERVENTIONS:
Diagnostic Test: Coronariography — Patients were classified as MICAD or MINOCA by the presence or absence of an epicardial vessel with ≥50% stenosis after performing a coronariography.

SUMMARY:
Around 10% of patients with myocardial infarction (MI) present with nonobstructive coronary arteries (MINOCA) which pathophysiology is often uncertain. The aim of the study is to evaluate inflammation and endothelial dysfunction biomarkers in MINOCA patients during both acute and stable phases, comparing them with those with MI and obstructive coronary arteries (MICAD).

DETAILED DESCRIPTION:
Prospective observational study in patients with Myocardial Infarction (MI) divided into two groups: MI with obstructive coronary arteries (MICAD) and MI with non-obstructive coronary arteries (MINOCA). Levels of interleukin-6, tumor necrosis factor-alpha, high-sensitivity C- reactive protein, and asymmetric dimethylarginine will be determined at three time points: within the 24 hours from the onset of pain, discharge, and two months after MI. The association of biomarkers, normalized by peak troponin value, with the risk of MINOCA will be evaluated using logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with Myocardial Infarction and undergo a coronariography
* Patients must sign informed consent.

Exclusion Criteria:

* Patients who don´t sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years old admitted to our hospital with Myocardial Infarction and undergo a coronariography.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Levels of interleukin-6 (pg/ml) and tumor necrosis factor-alpha (pg/ml) | At three time points: within the 24 hours from the onset of pain, on the 5th day of admission, and two months after MI.
  Levels of interleukin-6 (pg/ml) and tumor necrosis factor-alpha (pg/ml) will be determined.
Levels of endhotelial disfunction biomarkers | At three time points: within the 24 hours from the onset of pain, on the 5th day of admission, and two months after MI.
  Levels of asymmetric dimethylarginine will be determined
Levels of high-sensitivity C-reactive protein (mg/L) | t three time points: within the 24 hours from the onset of pain, on the 5th day of admission, and two months after MI.
  Levels of high-sensitivity C-reactive protein (mg/L) will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Getafe, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No